CLINICAL TRIAL: NCT06534697
Title: Analgesic Efficacy of Fascia Iliaca Block for Postoperative Pain Control After Elective Hip Arthroplasty: a Randomised Controlled Study
Brief Title: Fascia Iliaca Block for Postoperative Pain Control After Elective Hip Arthroplasty
Acronym: FIB-PAIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foisor Orthopedics Clinical Hospital (Other)
Responsible Party: Principal Investigator, Anastase Denisa, Consultant of anesthesiology and Intensive Care, Foisor Orthopedics Clinical Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07062024
Record Dates: First submitted 2024-07-25; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Hip Osteoarthritis
Keywords: Fascia iliaca block; Postoperative pain
MeSH Terms: conditions — Osteoarthritis, Hip; Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride; Glucose; Water

STUDY DESIGN:
Intervention Model Description: All enrolled patients will receive spinal anesthesia and preoperatively FIB for analgesia. The investigators randomly define three patient groups using the envelope method: Group 1, receiving 40 ml naropin 0,25% in saline; Group 2, receiving 40 ml naropin 0,25% in dextrose 5%; and Group 3, receiving 40 ml dextrose 10%. After the regression of spinal anesthesia, all the patients receive the same multimodal pain therapy according to the visual analog scale (VAS), including Paracetamol IV, NSAID, and morphine, according to the pain protocol in our hospital. The administration of morphine is according to our hospital protocol. The primary endpoint of the study is total morphine (mg) consumption at 24 hours postoperatively, and the second goal was length of stay and the risk of falls.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Naropin 0.25% in sodium chloride (Active Comparator): Preoperative supra inguinal fascia iliaca block with 40 ml naropin 0,25% in sodium chloride.
  Interventions: Drug: Naropin, 0.2% Injectable Solution in Sodium chloride
- Naropin 0.25% in dextrose 5% (Active Comparator): Preoperative supra inguinal fascia iliaca block with 40 ml naropin 0,25% in dextrose 5%.
  Interventions: Drug: Naropin, 0.2% Injectable Solution in dextrose 5%
- Placebo (Placebo Comparator): Preoperative supra inguinal fascia iliaca block with 40 ml dextrose 10%.
  Interventions: Drug: Dextrose 10 % in Water

INTERVENTIONS:
Drug: Naropin, 0.2% Injectable Solution in Sodium chloride — Preoperative fascia iliaca block with 40 ml volume of naropin 0,25% in sodium chloride
  Other Names: Ropivacaine 0.25%-Sodium chloride
  Arms: Naropin 0.25% in sodium chloride
Drug: Naropin, 0.2% Injectable Solution in dextrose 5% — Preoperative fascia iliaca block with 40 ml volume of naropin 0,25% in dextrose 5%
  Other Names: Ropivacaine 0.25%-Dextrose 5%
  Arms: Naropin 0.25% in dextrose 5%
Drug: Dextrose 10 % in Water — Preoperative fascia iliaca block with 40 ml volume of dextrose 10%
  Other Names: Dextrose 10%
  Arms: Placebo

SUMMARY:
This clinical trial aims to assess the analgesic efficacy of ultrasound-guided FIB using different analgesic combinations administered into the iliac fascia compartment. The main question it aims to answer is:

·What is the total morphine (mg) consumption at 24 hours postoperatively for each of the three groups?

The secondary questions are:

* What is the length of stay in hospital for each group?
* What is the risk of falling associated with the use of fascia iliaca block? Researchers will compare two analgesic combinations of local anesthestic naropin 0,25% versus dextrose 10% administered by fascia iliaca block for postoperative pain after total hip arthroplasty.

DETAILED DESCRIPTION:
The investigators plan to conduct a single-center, prospective, blinded, randomized controlled study of 150 eligible patients undergoing elective THA via a miniinvasive anterior approach starting June 2024. All patients will receive spinal anesthesia and preoperatively FIB for analgesia. The investigators define randomly three patient groups: Group 1, receiving 40 ml naropin 0,25% in saline, Group 2, receiving 40 ml naropin 0,25% in dextrose 5%, and Group 3, receiving 40 ml dextrose 10%. After the regression of spinal anesthesia, all the patients receive the same multimodal pain therapy according to the visual analog scale (VAS), including Paracetamol IV, NSAID, and morphine, according to the pain protocol in our hospital. The primary endpoint of the study is total morphine (mg) consumption at 24 hours postoperatively, and the secondary goals were length of stay and the risk of fall.

ELIGIBILITY:
Inclusion Criteria:

* Indication of total primary hip arthroplasty
* ASA I-III
* BMI<40 kg/m2

Exclusion Criteria:

* Inability or refusal to sign informed consent
* Known allergies to any of the drugs used in the study
* Hepatic or renal insufficiency
* Gastritis or gastroduodenal ulcer
* Opioid dependency
* Coagulopathy
* Pregnancy
* Scars in the surgery and fascia iliaca block areas
* Clinical evidence of peripheral neuropathies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-07-22 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
The total morphine consumption | 24 hours postoperatively
  The total morphine consumption is measured in mg

SECONDARY OUTCOMES:
The risk of fall | Up to 1 week
  The percent of the number of falls reported to the number of the patients for each arm
Length of stay in hospital | Up to 1 week
  The duration between admision and discharge of the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Denisa Anastase, MD, PhD, Principal Investigator — Foisor OCH; Simona Anastase, MD, PhD, Study Director — Foisor OCH

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Desmet M, Vermeylen K, Van Herreweghe I, Carlier L, Soetens F, Lambrecht S, Croes K, Pottel H, Van de Velde M. A Longitudinal Supra-Inguinal Fascia Iliaca Compartment Block Reduces Morphine Consumption After Total Hip Arthroplasty. Reg Anesth Pain Med. 2017 May/Jun;42(3):327-333. doi: 10.1097/AAP.0000000000000543. PMID 28059869
- [Background] Shariat AN, Hadzic A, Xu D, Shastri U, Kwofie K, Gandhi K, McCally CM, Gratenstein K, Vandepitte C, Gadsden J, Unis D. Fascia lliaca block for analgesia after hip arthroplasty: a randomized double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2013 May-Jun;38(3):201-5. doi: 10.1097/AAP.0b013e31828a3c7c. PMID 23558369
- [Background] Wee TC, Neo EJR, Tan YL. Dextrose prolotherapy in knee osteoarthritis: A systematic review and meta-analysis. J Clin Orthop Trauma. 2021 May 20;19:108-117. doi: 10.1016/j.jcot.2021.05.015. eCollection 2021 Aug. PMID 34046305
- [Background] Cui X, Cheng Z, Zhang T, Xu H, Luan H, Feng J, Zhang X, Zhu P. Effect of pericapsular nerve group block and suprainguinal fascia iliaca block on postoperative analgesia and stress response in elderly patients undergoing hip arthroplasty: a prospective randomized controlled double-blind trial. BMC Anesthesiol. 2024 Jul 2;24(1):220. doi: 10.1186/s12871-024-02604-8. PMID 38956469